CLINICAL TRIAL: NCT05676879
Title: The Effect of Ice Massage Applied to SP6 Point on Labor Pain, Labor Comfort, Labor Duration, and Anxiety
Brief Title: Ice Massage Applied to SP6 Point at Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Hülya TÜRKMEN, associate professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BalıkesirK
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Labor Pain; Labor Comfort; Duration of Labor; Anxiety
Keywords: Labor Pain; SP6 Acupoint; Labor comfort; duration of labor; anxiety
MeSH Terms: conditions — Labor Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Ice massage was applied to the SP6 points (SP6 point is located 3-4 fingers above the posterior malleolus bone, that is, 4 fingers above the ankle) of the pregnant women in first stage of childbirth at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilatations during 3 contractions. In order to prevent direct contact of ice with the skin, ice was applied as ice cubes wrapped in gauze.
  Interventions: Other: Ice massage was applied to the SP6 points
- Control Group (No Intervention): All the pregnant women, those in the control group, were provided with standard midwifery care.

INTERVENTIONS:
Other: Ice massage was applied to the SP6 points — Ice massage was applied to the SP6 points (SP6 point is located 3-4 fingers above the posterior malleolus bone, that is, 4 fingers above the ankle) of the pregnant women in first stage of childbirth at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilatations during 3 contractions.
  Arms: Intervention Group

SUMMARY:
Purpose: In the study , it was aimed to determine the effect of ice massage applied to SP6 point during labor on labor pain, labor comfort, labor duration, and anxiety.

Design: A single blind, randomized controlled experimental trial Setting and Participants: 100 primiparas, 50 in the intervention group and 50 in the control group, with 4-5 cm cervical dilatations were included in the study. Ice massage was applied to the SP6 point of the pregnant women in the intervention group at 4-5 cm, 6-7 cm, and 8-9 cm dilatations during three contractions.

Measurement Tools: The Pregnant Information Form, VAS, the Partograph Form, Childbirth Comfort Questionnaire (CCQ), and the State Anxiety Scale were used to collect data.

DETAILED DESCRIPTION:
The study was conducted as a randomized controlled trial in the Delivery Room of Ataturk City Hospital located in Balikesir province of Turkey between December 2021 and July 2022.

Participants The study sample size was calculated by using G*Power 3 power calculations based on previous studies in which ice massage was applied to acupressure points during labor. Impact estimation was obtained from the findings of the study conducted by Hajiamini et al., who reported pain severity as 5.90 ± 1.84 in the ice massage group and 7.10 ± 1.64 in the control group 30 minutes after the ice massage application. In the present study, it was aimed to determine a similar difference. The sample size for each group was determined to be at least 47 individuals. Accordingly, 50 primiparas were assigned to the intervention group and the control group each. The power analysis performed showed that the sample size of the study had a power as α = 0.05, Power = 0.91, df = 98. The decrease observed in labor pain at 4-5 cm cervical dilatation compared to the control group had an impact size of 0.61.

The inclusion criteria for the primiparas were having a single healthy fetus, having a gestational age between 38 and 40 weeks, expecting vaginal delivery, having fetal cephalic presentation, having no chronic diseases, not having a high-risk pregnancy, being in stage 1 of childbirth, and having a 4-5 cm cervical dilatation. Pregnant women who were multiparous, had multiple pregnancies, had high-risk pregnancy, had delivery with complications, and came to the clinic after 4-5 cm dilatation were excluded from the study.

Single blind block randomization for pregnant women who met the inclusion criteria was achieved by using Sequence Generator method located under the subheading of Numbers at random.org website. In the program, two columns were created according to the sample size. The pregnant women were randomly assigned to Column 1 or Column 2 according to their registration number. The assignment of the columns to either the intervention group or the control group was done through a draw. Ice massage was applied to SP6 points of the pregnant women in the intervention group, while the pregnant women in the control group was provided with standard midwifery care.

Data collection The Pregnant Information Form (PIF), Visual Analog Scale (VAS-1), and Childbirth Comfort Questionnaire (CCQ) were administered to the pregnant women who were at stage 1 of delivery and 4-5 cm cervical dilatation. Each group was provided with standard midwifery care, and intervention was made to the women in the intervention group at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilatation during three contractions. Immediately after the interventions, VAS-2, VAS-3, and VAS-4 were applied. In addition, following the intervention made at 6-7 cm cervical dilatation, The State Anxiety Scale (STAI-I) was applied between the contractions. After the interventions were completed, CCQ was applied again at 8-9 cm cervical dilatation. The pregnant women in the control group were administered VAS-2, VAS-3, and VAS-4 at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilatations, STAI-I at 6-7 cm cervical dilatation, and CCQ at 8-9 cm cervical dilatation.

Measurement tools The study data were collected through The Pregnant Information Form, VAS, Partograph Form, Childbirth Comfort Scale, and the State Anxiety Scale.

The Pregnant Information Form (PIF): The form consists of 22 questions inquiring about the sociodemographic, gynecological, and obstetric characteristics of the pregnant women.

Visual Analog Scale (VAS): The scale was used in order to measure labor pain. It is made up of a vertical line ranging from 0 to 10. In the study, VAS was applied before the intervention at 4-5 cm cervical dilatation (VAS-I) and after the intervention at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilatations (VAS-2, VAS-3, VAS-4, respectively).

Childbirth Comfort Questionnaire (CCQ): The 9-item scale is a 5-point Likert type scale (1=Absolutely Disagree, 5=Absolutely Agree). The score to be obtained from the scale ranges between 9-45. A high score indicates a high level of comfort. In the present study, this value for the scale was determined to be 0.72. CCQ was applied two times in the study, once at 4-5 cm cervical dilatation before the intervention and once at 8-9 cm dilatation after the intervention.

State Anxiety Scale (STAI-I): The 4-point Likert type scale (1=Almost Never, 4=Almost Always) consists of 20 questions. There are two types of statements on the scale. Direct statements express negative emotions, while reverse statements express positive emotions. Weighted total score is calculated for both direct and reverse statements. The totals score obtained from negative statements is subtracted from the total score obtained from positive statements. A pre-determined constant number (50) is added to this number obtained. The final score obtained is the individual's anxiety score. The scores obtained from the scale varies between 20 and 80. A high score shows a high level of anxiety.

Intervention Ice massage was applied to the SP6 points (SP6 point is located 3-4 fingers above the posterior malleolus bone, that is, 4 fingers above the ankle) of the pregnant women in first stage of childbirth at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilatations during 3 contractions. In order to prevent direct contact of ice with the skin, ice was applied as ice cubes wrapped in gauze. Standard midwifery care was provided to the women in both groups. In the hospital where the study was conducted, cervical dilatation and effacement follow-up, contraction and fetal heart rate follow-up, vital signs monitoring, and routine oxytocin induction are applied as standard midwifery care. In addition, pregnant women are provided with information on breathing and pushing techniques. 4 drop/min 10IU/ml oxytocin induction was applied to all pregnant women in both groups at 4-5 cm cervical dilatation. Oxytocin induction was increased by 4 drops at every 20 minutes. It was applied at a maximum dose of 40 drop/min.

ELIGIBILITY:
Inclusion Criteria:

* expected vaginal delivery
* single healthy fetus
* primipara
* in the first phase of the labor

Exclusion Criteria:

* multipara
* risky pregnancy
* child with complications
* multiple pregnancies
* premature delivery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
severity of labor pain by VAS | immediately after the intervention
  The scale was used in order to measure labor pain. It is made up of a vertical line ranging from 0 to 10 (Ferreira-Valente et al., 2011). In the study, VAS was applied before the intervention at 4-5 cm cervical dilatation (VAS-I) and after the intervention at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilatations (VAS-2, VAS-3, VAS-4, respectively).

SECONDARY OUTCOMES:
duration of labor | during the procedure
  duration of active phase and transition phase of labor (4-10cm cervical dilatation)

CONTACTS AND LOCATIONS:
Locations (1):
- Hülya Türkmen, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No